CLINICAL TRIAL: NCT02960217
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Crossover Study to Assess the Efficacy and Safety of UX007 in the Treatment of Movement Disorders Associated With Glucose Transporter Type 1 Deficiency Syndrome (Glut1 DS)
Brief Title: Crossover Study to Assess the Efficacy and Safety of UX007 in the Treatment of Movement Disorders Associated With Glucose Transporter Type 1 Deficiency Syndrome (Glut1 DS)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was halted prematurely due to lack of efficacy.
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UX007G-CL301
Expanded Access: NCT03773770 (Available)
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Glucose Transporter Type 1 Deficiency Syndrome (Glut1 DS)
MeSH Terms: conditions — Glut1 Deficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Double-Blind UX007 Followed by Placebo (Experimental): Participants will first receive UX007 (dosed according to an age- and weight-based strategy, up to a maximum daily administration of 130 g) for 10 weeks. After a washout period of 2 weeks, they will then receive placebo for 10 weeks.
  Participants will have the option of rolling into the open label Extension Period, to continue UX007 treatment for up to 3 years.
  Interventions: Drug: UX007; Drug: Placebo
- Double Blind Placebo Followed by UX007 (Experimental): Participants will first receive Placebo for 10 weeks. After a washout period of 2 weeks, they will then receive UX007 (dosed according to an age- and weight-based strategy, up to a maximum daily administration of 130 g) for 10 weeks.
  Participants will have the option of rolling into the open label Extension Period, to continue UX007 treatment for up to 3 years.
  Interventions: Drug: UX007; Drug: Placebo

INTERVENTIONS:
Drug: UX007 — liquid for oral (PO) administration
Drug: Placebo — liquid safflower oil for PO administration

SUMMARY:
The primary objective of the study was to evaluate the efficacy and safety of UX007 in the treatment of disabling paroxysmal movement disorders associated with Glut1 DS.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Glut1 DS confirmed by SLC2A1 mutation
2. Males and females, aged ≥6 years old at the time of informed consent
3. At least 8 disabling paroxysmal movement disorder events in the 12 weeks prior to the Screening, by subject or caregiver report or At least 6 disabling paroxysmal movement disorder events in any 6 consecutive week period, over the last 12 week period prior to the Screening, by subject or caregiver report
4. At least 4 disabling paroxysmal movement disorder events in 6 week Run-in Period, reported in the daily electronic Glut1 DS symptom diary
5. ≥80% compliance with daily electronic Glut1 DS symptom diary completion during the Run in Period
6. Not on ketogenic diet (KD), modified KD, or ketosis-inducing modified-fat diet for at least 3 months prior to Screening
7. Plasma level of beta-hydroxybutyrate (BHB) ≤ 1 mmol/L (non-fasting) at Screening
8. Provide written or verbal assent (if possible) and written informed consent by the patient(if an adult), or by a legally authorized representative after the nature of the study has been explained, and prior to any research-related procedures
9. Must, in the opinion of the Investigator, be willing and able to complete key aspects of the study and be likely to complete the 22-week, placebo-controlled, treatment period
10. Patient (or caregiver) must, in the opinion of the Investigator, be able to comply with accurate completion of the study daily electronic Glut1 DS symptom diary
11. Females of child-bearing potential must have a negative urine pregnancy test at Screening and Baseline and be willing to have additional pregnancy tests during the study. Females considered not to be of child-bearing potential include those who have not experienced menarche, are post-menopausal (defined as having no menses for at least 12 months without an alternative medical cause) or are permanently sterile due to total hysterectomy, bilateral salpingectomy, or bilateral oophorectomy.
12. Participants of child-bearing potential or fertile males with partners of child-bearing potential who are sexually active must consent to use a highly effective method of contraception as determined by the site Investigator from the period following the signing of the informed consent through 30 days after last dose of study drug

Exclusion Criteria:

1. Any known hypersensitivity to triheptanoin or safflower oil that, in the judgment of the Investigator, places the subject at increased risk for adverse effects
2. Prior use of triheptanoin within 30 days prior to Screening
3. History of, or current suicidal ideation, behavior and/or attempts per Columbia Suicide Severity Rating Scale (C-SSRS) at Screening or Baseline
4. Pregnant and/or breastfeeding an infant at Screening or Baseline
5. Participants unwilling or unable to discontinue use of a prohibited medication or other substance that may confound study objectives (medium chain triglyceride [MCT] oil, barbiturates, pancreatic lipase inhibitors, KetoCal or other KD supplements, and/or KD])
6. Glut1 DS treatment regimen, including antiepileptic drugs (AEDs), should be stable for at least 30 days prior to Screening
7. Use of any investigational product (drug, medical food, or supplement, including MCT oil, including coconut oil) within 30 days prior to Screening
8. Has a concurrent disease or condition, or laboratory abnormality that, in the view of the Investigator, places the subject at high risk of poor treatment compliance or of not completing the study, or would interfere with study participation or introduces additional safety concerns
9. Feeding or nutrition that, in the opinion of the dietitian, potentially affects consistent administration of study drug

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (12):
- United States (4):
  - Colorado Children's Hospital, Aurora, Colorado
  - Nicklaus Children's Hospital, Miami, Florida
  - Center for Rare Neurological Diseases, Norcross, Georgia
  - Columbia University Medical Center, New York, New York
- Hopital Robert Debre, Paris, France
- Germany (3):
  - University of Essen, Essen
  - Klinikum der Universitat München, München
  - Universitaetklinikum Tuebingen, Tübingen
- IRCCS Fondazione Istituto Neurologico Nazionale C. Mondino, Pavia, Italy
- Hospital Vall d'Hebron, Barcelona, Spain
- United Kingdom (2):
  - Leonard Wolfson Experimental Neurology Centre, London
  - Sheffield Children's NHS Foundation Trust, Sheffield

REFERENCES:
- See also: Company Website — http://www.ultragenyx.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During a 6-week Run-in Period, participants recorded disabling paroxysmal movement disorder events in a daily electronic Glut1 DS movement disorder diary.
  One participant was randomized but did not receive any treatment due to a protocol violation; this participant was not included in any analysis population.
Groups:
- Double-Blind UX007 Followed by Placebo: Double-Blind Maintenance Phase: Participants received UX007 (dosed according to an age- and weight-based strategy, up to a maximum daily administration of 130 g) for 10 weeks. After a washout period of 2 weeks, they then received placebo for 10 weeks.
  Participants had the option of rolling into the Open-Label Extension Phase, to continue UX007 treatment (dosed according to an age- and weight-based strategy, up to a maximum daily administration of 130 g) for up to 3 years.
- Double-Blind Placebo Followed by UX007: Double-Blind Maintenance Phase: Participants received placebo for 10 weeks. After a washout period of 2 weeks, they then received UX007 (dosed according to an age- and weight-based strategy, up to a maximum daily administration of 130 g) for 10 weeks.
  Participants had the option of rolling into the Open-Label Extension Phase, to continue UX007 treatment (dosed according to an age- and weight-based strategy, up to a maximum daily administration of 130 g) for up to 3 years.
Period: Maintenance Phase: Treatment Period 1
Arm/Group | Double-Blind UX007 Followed by Placebo | Double-Blind Placebo Followed by UX007
Started (Randomized and treated) | 22 | 21
Completed | 21 | 21
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Maintenance Phase: Crossover Washout
Arm/Group | Double-Blind UX007 Followed by Placebo | Double-Blind Placebo Followed by UX007
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0
Period: Maintenance Phase: Treatment Period 2
Arm/Group | Double-Blind UX007 Followed by Placebo | Double-Blind Placebo Followed by UX007
Started | 21 | 21
Completed | 20 | 18
Not Completed | 1 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Other, Not Specified | 0 | 1
Period: Open-Label Extension Phase
Arm/Group | Double-Blind UX007 Followed by Placebo | Double-Blind Placebo Followed by UX007
Started | 20 | 13 (5 participants completed the double blind period but did not continue in the open label period.)
Completed | 0 | 0
Not Completed | 20 | 13
Not completed — Adverse Event | 1 | 0
Not completed — Sponsor Decision | 18 | 11
Not completed — Lack of Efficacy | 1 | 1
Not completed — Other, Not Specified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug.
Groups:
- Double-Blind UX007 Followed by Placebo: Double-Blind Maintenance Period: Participants received UX007 (dosed according to an age- and weight-based strategy, up to a maximum daily administration of 130 g) for 10 weeks. After a washout period of 2 weeks, they then received placebo for 10 weeks.
  Participants had the option of rolling into the Open-Label Extension Period, to continue UX007 treatment for up to 3 years.
- Double-Blind Placebo Followed by UX007: Double-Blind Maintenance Period: Participants received placebo for 10 weeks. After a washout period of 2 weeks, they then received UX007 (dosed according to an age- and weight-based strategy, up to a maximum daily administration of 130 g) for 10 weeks.
  Participants had the option of rolling into the Open-Label Extension Period, to continue UX007 treatment for up to 3 years.
- Total: Total of all reporting groups
Arm/Group | Double-Blind UX007 Followed by Placebo | Double-Blind Placebo Followed by UX007 | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.41 (13.156) | 18.37 (5.730) | 20.95 (10.425)
Age, Customized [Count of Participants; unit: Participants]
  < 18 years old | 7 | 9 | 16
  >/= 18 years old | 15 | 12 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 10 | 9 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 17 | 17 | 34
  Unknown or Not Reported | 4 | 4 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 1 | 1
  White | 18 | 16 | 34
  Missing | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Maintenance Phase Movement Disorder Frequency
Description: The frequency of paroxysmal movement disorders captured as disabling movement disorder events (normalized to a 4-week rate) observed during the Maintenance Phase in participants treated with UX007 versus placebo, as recorded by the subject/caregiver in an event-based daily Glut1 DS symptom diary.
Time Frame: Maintenance Phase (up to Week 22)
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: movement disorder events per 4 weeks
Groups:
- Double-Blind UX007: UX007 (dosed according to an age- and weight-based strategy, up to a maximum daily administration of 130 g) for 10 weeks.
- Double-Blind Placebo: Placebo for 10 weeks.
Arm/Group | Double-Blind UX007 | Double-Blind Placebo
Number analyzed (Participants) | 43 | 42
movement disorder events per 4 weeks | 14.26 [0.0 to 112.0] | 11.81 [0.5 to 112.0]
Statistical Analysis 1: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Participants completing both UX007 treatment period and placebo period (n=42). Per protocol, when the normality assumption is not met (p value for Wilk-Shapiro test < 0.05), Wilcoxon rank-sum test will be considered as the primary analysis to assess treatment difference in movement disorder event frequency; Test type: Superiority; p = 0.2684, Wilcoxon Rank Sum test — Hodges-Lehmann estimate of the location shift with 95% confidence interval (CI) and Wilcoxon Rank Sum test p-value are based on Wilcoxon rank-sum test; Hodges-Lehmann estimate (Median Diff.) = 1.46, 95% CI 2-sided [-1.12 to 4.36]
Statistical Analysis 2: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p < 0.0001, Wilk-Shapiro test for normality

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, and Discontinuations Due to TEAEs
Description: An Adverse Event (AE) was defined as any untoward medical occurrence, whether or not considered drug related. Serious adverse events (SAE) was defined as an AE that at any dose, in the view of either the Investigator or Ultragenyx, results in any of the following outcomes: death; a life-threatening AE; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant incapacity or disability (substantial disruption of the ability to conduct normal life functions); a congenital anomaly/birth defect; other important medical event. All reported AEs with with a start date that occurred or worsened in severity on or after the first dose of study drug in the corresponding treatment period and before the first dose of study drug in the next treatment period were defined as TEAEs. AEs were graded as 1=mild, 2=moderate, 3=severe, 4=life=threatening, 5=death.
Time Frame: From first dose of study drug through 30-35 days after final dose. Mean (SD) treatment duration was 65.7 (12.06) and 68.3 (7.04) days for double-blind UX007 and placebo, and 305.0 (122.71) days for open-label UX007.
Population: Safety Analysis Set: all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Double-Blind UX007: Double-Blind Maintenance Phase: Participants received UX007 (dosed according to an age- and weight-based strategy, up to a maximum daily administration of 130 g) for 10 weeks.
- Double-Blind Placebo: Double-Blind Maintenance Phase: Participants received placebo for 10 weeks.
- Open-Label UX007: Open-Label Extension Phase: Participants continued UX007 treatment for up to 3 years.
Arm/Group | Double-Blind UX007 | Double-Blind Placebo | Open-Label UX007
Number analyzed (Participants) | 43 | 42 | 33
Participants
  TEAEs | 40 | 34 | 28
  Serious TEAEs | 2 | 1 | 2
  Treatment-Related TEAEs | 33 | 19 | 17
  Treatment-Related Serious TEAEs | 1 | 0 | 0
  Grade 3 or 4 TEAEs | 4 | 3 | 3
  Grade 4 TEAEs | 0 | 0 | 0
  Gastrointestinal TEAEs | 32 | 17 | 18
  TEAEs Leading to Treatment Discontinuation | 2 | 1 | 0
  TEAEs Leading to Study Discontinuation | 2 | 1 | 0
  TEAEs Leading to Death | 0 | 0 | 0

3. Primary Outcome: Baseline and Post-Baseline Columbia Suicide Severity Rating Scale (C-SSRS) Responses During Double-Blind Treatment Period
Description: The C-SSRS is a participant-rated questionnaire to assess suicidal ideation, suicidal behavior, and self-injurious behavior with no suicidal intent (yes or no responses). Positive responses (i.e., 'Yes') to C-SSRS questions correspond to events in these categories with the exception of the category 'No events'. Suicidal ideation includes the following subcategories: passive; active-nonspecific; active-method/no intent/no plan; active-intent/with or without method/no plan; active-method/intent/plan. Suicidal behavior includes the following subcategories: suicide attempt; interrupted attempt; aborted attempt; preparatory actions toward immanent suicidal behaviors; completed suicide. Suicidal ideation and/or suicidal behavior category includes participants with positive responses in the category suicidal ideation and/or suicidal behavior.
Time Frame: Baseline, up to Week 22
Population: Safety Analysis Set: all randomized participants who received at least 1 dose of study drug. Participants with a baseline (BL) and postbaseline (PB) assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind UX007 | Double-Blind Placebo
Number analyzed (Participants) | 40 | 40
Participants
  BL: No Events | 38 | 38
  PB: No Events | 40 | 39
  BL: Suicidal Ideation | 1 | 1
  PB: Suicidal Ideation | 0 | 0
  BL: Suicidal Behavior | 1 | 1
  PB: Suicidal Behavior | 0 | 1
  BL: Suicidal Ideation and/or Behavior | 2 | 2
  PB: Suicidal Ideation and/or Behavior | 0 | 1
  BL: Self-Injurious Behavior, No Suicidal Intent | 1 | 1
  PB: Self-Injurious Behavior, No Suicidal Intent | 0 | 1

4. Secondary Outcome: Change From Period Baseline in 12 Minute Walk Test (12MWT) Distance at Treatment Week 10
Description: Walking capacity and endurance, as determined by the distance in meters walked in 12 minutes during the 12MWT.
Time Frame: Period Baseline (defined as the last non-missing assessment prior to or on the date of the first dose of study drug for each double-blind Treatment Period), Week 10
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug. Participants who had an assessment.
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | Double-Blind UX007 | Double-Blind Placebo
Number analyzed (Participants) | 36 | 38
meters | -15.9 (25.63) | -33.0 (24.91)
Statistical Analysis 1: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Number of participants in this analysis completed both UX007 treatment period and placebo treatment period (n=34); Test type: Superiority; p = 0.6419, Wilcoxon Rank Sum test — Hodges-Lehmann estimate of the location shift with 95% CI and Wilcoxon Rank Sum test p-value are based on Wilcoxon rank-sum test; Hodges-Lehmann estimate (Median Diff.) = 25.00, 95% CI 2-sided [-62.5 to 91.5]
Statistical Analysis 2: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.0005, Wilk-Shapiro Test for Normality

5. Secondary Outcome: Change From Period Baseline in Patient Reported Outcomes Measurement Information System (PROMIS) Health Assessment Questionnaire (Adult Form) Physical Function Score at Treatment Week 10
Description: The PROMIS was developed by the National Institutes of Health and uses domain-specific measures to assess patient well-being (Broderick et al. 2013; NIH 2015). It uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. For the Physical Function Mobility Domain, increases in score indicate greater mobility.
Time Frame: as for outcome 4
Population: Full Analysis Set: all randomized adult participants who received at least 1 dose of study drug. Participants who had an assessment.
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Double-Blind UX007 | Double-Blind Placebo
Number analyzed (Participants) | 23 | 25
T-score | -0.9 (0.67) | -0.9 (0.65)
Statistical Analysis 1: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.9513, ANCOVA — Based on an ANCOVA model including covariate for period baseline value, fixed effects for treatment sequence, treatment group, period, and a random effect for participant within the sequence; LS Mean Difference = -0.1, 95% CI 2-sided [-2.0 to 1.9], Standard Error of Mean 0.91
Statistical Analysis 2: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.8214, Wilk-Shapiro Test for Normality

6. Secondary Outcome: Change From Period Baseline in PROMIS Health Assessment Questionnaire (Adult Form) Fatigue Score at Treatment Week 10
Description: The PROMIS was developed by the National Institutes of Health and uses domain-specific measures to assess patient well-being (Broderick et al. 2013; NIH 2015). It uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. For the Fatigue Domain, decreases in score indicate less fatigue.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Double-Blind UX007 | Double-Blind Placebo
Number analyzed (Participants) | 23 | 25
T-score | 2.9 (1.40) | 0.9 (1.36)
Statistical Analysis 1: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.1572, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = 2.0, 95% CI 2-sided [-0.8 to 4.7], Standard Error of Mean 1.32
Statistical Analysis 2: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.8451, Wilk-Shapiro Test for Normality

7. Secondary Outcome: Change From Period Baseline in PROMIS Health Assessment Questionnaire (Adult Form) Sleep Disturbance Score at Treatment Week 10
Description: The PROMIS was developed by the National Institutes of Health and uses domain-specific measures to assess patient well-being (Broderick et al. 2013; NIH 2015). It uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. For the Sleep Disturbance Domain, decreases in score indicate less sleep disturbance.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Double-Blind UX007 | Double-Blind Placebo
Number analyzed (Participants) | 23 | 25
T-score | 0.4 (1.24) | 0.7 (1.20)
Statistical Analysis 1: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.8345, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-3.8 to 3.1], Standard Error of Mean 1.66
Statistical Analysis 2: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.2894, Wilk-Shapiro Test for Normality

8. Secondary Outcome: Change From Period Baseline in PROMIS Health Assessment Questionnaire (Adult Form) Pain Interference Score at Treatment Week 10
Description: The PROMIS was developed by the National Institutes of Health and uses domain-specific measures to assess patient well-being (Broderick et al. 2013; NIH 2015). It uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. For the Pain Interference Domain, decreases in scores indicate less pain interference.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Double-Blind UX007 | Double-Blind Placebo
Number analyzed (Participants) | 23 | 25
T-score | 4.5 (1.64) | 3.7 (1.58)
Statistical Analysis 1: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.0005, Wilk-Shapiro Test for Normality
Statistical Analysis 2: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Number of participants in this analysis completed both UX007 treatment period and placebo treatment period (n=21); Test type: Superiority; p = 0.4898, Wilcoxon Rank Sum test — [p-value comment as in outcome 4, analysis 1]; Hodges-Lehmann estimate (Median Diff.) = 0.2, 95% CI 2-sided [-5.4 to 5.8]

9. Secondary Outcome: Change From Period Baseline in PROMIS Health Assessment Questionnaire (Adult Form) Cognitive Function Score at Treatment Week 10
Description: The PROMIS was developed by the National Institutes of Health and uses domain-specific measures to assess patient well-being (Broderick et al. 2013; NIH 2015). It uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. The Cognitive Function Domain measures cognitive function impairment. Decreases in score indicate less cognitive function impairment.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Double-Blind UX007 | Double-Blind Placebo
Number analyzed (Participants) | 23 | 25
T-score | 2.0 (1.29) | 1.2 (1.25)
Statistical Analysis 1: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.5853, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = 0.8, 95% CI 2-sided [-2.2 to 3.8], Standard Error of Mean 1.42
Statistical Analysis 2: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.1066, Wilk-Shapiro Test for Normality

10. Secondary Outcome: Change From Period Baseline in PROMIS Health Assessment Questionnaire (Adult Form) Social Roles and Activities Score at Treatment Week 10
Description: The PROMIS was developed by the National Institutes of Health and uses domain-specific measures to assess patient well-being (Broderick et al. 2013; NIH 2015). It uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. For the Social Roles and Activities Domain, decreases in score indicate worse /less or decrease of performance in social roles and activities.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Double-Blind UX007 | Double-Blind Placebo
Number analyzed (Participants) | 23 | 25
T-score | -4.1 (1.35) | -2.3 (1.32)
Statistical Analysis 1: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.1875, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -1.8, 95% CI 2-sided [-4.6 to 1.0], Standard Error of Mean 1.33
Statistical Analysis 2: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.2034, Wilk-Shapiro Test for Normality

11. Secondary Outcome: Change From Period Baseline in PROMIS Health Assessment Questionnaire (Adult Form) Anxiety Score at Treatment Week 10
Description: The PROMIS was developed by the National Institutes of Health and uses domain-specific measures to assess patient well-being (Broderick et al. 2013; NIH 2015). It uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. For the Anxiety Domain, decreases in scores indicate less anxiety.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Double-Blind UX007 | Double-Blind Placebo
Number analyzed (Participants) | 23 | 25
T-score | 3.1 (1.49) | 0.5 (1.45)
Statistical Analysis 1: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.1138, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = 2.6, 95% CI 2-sided [-0.7 to 5.9], Standard Error of Mean 1.56
Statistical Analysis 2: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.1478, Wilk-Shapiro Test for Normality

12. Secondary Outcome: Change From Period Baseline in PROMIS Health Assessment Questionnaire (Pediatric/Parent-Proxy Form) Mobility Score at Treatment Week 10
Description: The PROMIS was developed by the National Institutes of Health and uses domain-specific measures to assess patient well-being (Broderick et al. 2013; NIH 2015) via parent/proxy. It uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. For the Mobility Domain, decreases in score indicate less mobility.
Time Frame: as for outcome 4
Population: Full Analysis Set: all randomized pediatric participants who received at least 1 dose of study drug. Participants who had an assessment.
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Double-Blind UX007 | Double-Blind Placebo
Number analyzed (Participants) | 16 | 13
T-score | -1.0 (1.62) | 0.0 (1.73)
Statistical Analysis 1: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.5505, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -1.0, 95% CI 2-sided [-4.6 to 2.6], Standard Error of Mean 1.62
Statistical Analysis 2: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.4459, Wilk-Shapiro Test for Normality

13. Secondary Outcome: Change From Period Baseline in PROMIS Health Assessment Questionnaire (Pediatric/Parent-Proxy Form) Upper Extremity Score at Treatment Week 10
Description: The PROMIS was developed by the National Institutes of Health and uses domain-specific measures to assess patient well-being (Broderick et al. 2013; NIH 2015) via parent/proxy. It uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. For the Upper Extremity Domain, decreases in score indicate less upper extremity movement.
Time Frame: as for outcome 4
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Double-Blind UX007 | Double-Blind Placebo
Number analyzed (Participants) | 16 | 13
T-score | -0.4 (1.91) | 1.3 (2.11)
Statistical Analysis 1: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.5544, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -1.7, 95% CI 2-sided [-8.1 to 4.6], Standard Error of Mean 2.84
Statistical Analysis 2: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.1104, Wilk-Shapiro Test for Normality

14. Secondary Outcome: Change From Period Baseline in PROMIS Health Assessment Questionnaire (Pediatric/Parent-Proxy Form) Fatigue Score at Treatment Week 10
Description: The PROMIS was developed by the National Institutes of Health and uses domain-specific measures to assess patient well-being (Broderick et al. 2013; NIH 2015) via parent/proxy. It uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. For the Fatigue Domain, decreases in score indicate less fatigue.
Time Frame: as for outcome 4
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Double-Blind UX007 | Double-Blind Placebo
Number analyzed (Participants) | 16 | 13
T-score | -1.8 (2.40) | -0.6 (2.64)
Statistical Analysis 1: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.7145, ANCOVA; LS Mean Difference = -1.2, 95% CI 2-sided [-8.5 to 6.1], Standard Error of Mean 3.27
Statistical Analysis 2: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.8255, Wilk-Shapiro Test for Normality

15. Secondary Outcome: Change From Period Baseline in PROMIS Health Assessment Questionnaire (Pediatric/Parent-Proxy Form) Pain Interference Score at Treatment Week 10
Description: The PROMIS was developed by the National Institutes of Health and uses domain-specific measures to assess patient well-being (Broderick et al. 2013; NIH 2015) via parent/proxy. It uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. For the Pain Interference Domain, decreases in score indicate less pain interference.
Time Frame: as for outcome 4
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Double-Blind UX007 | Double-Blind Placebo
Number analyzed (Participants) | 16 | 13
T-score | 3.2 (1.84) | 1.6 (1.96)
Statistical Analysis 1: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.4176, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = 1.5, 95% CI 2-sided [-2.5 to 5.6], Standard Error of Mean 1.82
Statistical Analysis 2: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.6557, Wilk-Shapiro Test for Normality

16. Secondary Outcome: Change From Period Baseline in PROMIS Health Assessment Questionnaire (Pediatric/Parent-Proxy Form) Peer Relationships Score at Treatment Week 10
Description: The PROMIS was developed by the National Institutes of Health and uses domain-specific measures to assess patient well-being (Broderick et al. 2013; NIH 2015) via parent/proxy. It uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. For the Peer Relationships Domain, decreases in score indicate worse functioning in peer relationships.
Time Frame: as for outcome 4
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Double-Blind UX007 | Double-Blind Placebo
Number analyzed (Participants) | 16 | 13
T-score | 2.0 (1.57) | -0.0 (1.64)
Statistical Analysis 1: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.0935, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = 2.0, 95% CI 2-sided [-0.4 to 4.5], Standard Error of Mean 1.09
Statistical Analysis 2: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.7267, Wilk-Shapiro Test for Normality

17. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I) at Treatment Week 10
Description: Participant/caregiver global impression of change in clinical status using the CGI-I. The CGI-I is a 7-point scale that assesses how much the participant's condition has improved or worsened relative to a baseline state at the beginning of the intervention and rated as: 1=very much better; 2=much better; 3=a little better; 4=no change; 5=a little worse; 6=much worse; 7=very much worse.
Time Frame: Week 10
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Double-Blind UX007 | Double-Blind Placebo
Number analyzed (Participants) | 38 | 40
score on a scale | 3.5 (0.20) | 3.6 (0.20)
Statistical Analysis 1: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.8329, ANCOVA — Based on an ANCOVA model including covariate for study baseline CGI-S score, fixed effects for treatment sequence, treatment group, period, and a random effect for subject within the sequence; LS Mean Difference = -0.1, 95% CI 2-sided [-0.6 to 0.5], Standard Error of Mean 0.28
Statistical Analysis 2: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.2348, Wilk-Shapiro Test for Normality

18. Secondary Outcome: Duration of Movement Disorder Events During Maintenance Phase
Description: Duration of disabling paroxysmal movement disorder events observed during the Maintenance Period of treatment, as recorded by the subject/caregiver in an event-based daily electronic Glut1 DS symptom diary.
Time Frame: Maintenance Phase (up to 22 weeks)
Population: Full Analysis Set: all randomized participants (or parent/proxy) who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Double-Blind UX007 | Double-Blind Placebo
Number analyzed (Participants) | 43 | 42
hours | 0.9 (1.98) | 0.7 (1.53)

19. Secondary Outcome: Change From Period Baseline in Cambridge Neuropsychological Test Automated Battery (CANTAB), Spatial Span (SSP) Span Length Scores at Treatment Week 10
Description: Cognitive function as measured by the CANTAB. CANTAB measures neuropsychological function using a standardized, computerized battery of tests designed to assess visual memory, working memory, new learning and reaction time. SSP Span Length assesses the cognitive domain of sequential memory, with scores on a discrete, ordinal scale from 2 to 9; higher scores indicate better function.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind UX007 | Double-Blind Placebo
Number analyzed (Participants) | 13 | 14
units on a scale | 0.1 (0.31) | 0.6 (0.29)
Statistical Analysis 1: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.0315, Wilk-Shapiro Test for Normality
Statistical Analysis 2: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Number of participants in this analysis completed both UX007 treatment period and placebo treatment period (n=13); Test type: Superiority; p = 0.2425, Wilcoxon Rank Sum test — [p-value comment as in outcome 4, analysis 1]; Hodges-Lehmann estimate (Median Diff.) = -0.5, 95% CI 2-sided [-1.5 to 0.5]

20. Secondary Outcome: Change From Period Baseline in CANTAB, Spatial Working Memory Between Errors (SWMBE) Scores at Treatment Week 10
Description: CANTAB measures neuropsychological function using a standardized, computerized battery of tests designed to assess visual memory, working memory, new learning and reaction time. SWMBE assesses the cognitive domain of working memory, with scores on a discrete, ordinal scale from 0 to 360; lower scores indicate better function.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind UX007 | Double-Blind Placebo
Number analyzed (Participants) | 13 | 14
units on a scale | -0.2 (2.94) | 0.2 (2.83)
Statistical Analysis 1: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.0072, Wilk-Shapiro Test for Normality
Statistical Analysis 2: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Number of participants in this analysis completed both UX007 treatment period and placebo treatment period (n=12); Test type: Superiority; p = 1.0000, Wilcoxon Rank Sum test — [p-value comment as in outcome 4, analysis 1]; Hodges-Lehmann estimate (Median Diff.) = 0.0, 95% CI 2-sided [-14.5 to 13.5]

21. Secondary Outcome: Change From Period Baseline in CANTAB, Spatial Working Memory Strategy (SWMS) Scores at Treatment Week 10
Description: CANTAB measures neuropsychological function using a standardized, computerized battery of tests designed to assess visual memory, working memory, new learning and reaction time. SWMS assesses the cognitive domain of executive function/strategy, with scores on a discrete, ordinal scale from 4 to 28; lower scores indicate better function.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind UX007 | Double-Blind Placebo
Number analyzed (Participants) | 13 | 14
units on a scale | 0.6 (0.77) | -0.4 (0.74)
Statistical Analysis 1: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.1076, ANCOVA — Based on an ANCOVA model including covariate for period baseline value, fixed effects for treatment sequence, treatment group, period, and a random effect for subject within the sequence; LS Mean Difference = 1.0, 95% CI 2-sided [-0.3 to 2.2], Standard Error of Mean 0.54
Statistical Analysis 2: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.7698, Wilk-Shapiro Test for Normality

22. Secondary Outcome: Change From Baseline in CANTAB, Paired Associates Learning Total Errors (PALTEA) at Treatment Week 10
Description: CANTAB measures neuropsychological function using a standardized, computerized battery of tests designed to assess visual memory, working memory, new learning and reaction time. PALTEA assesses the cognitive domain of episodic memory/new learning, with scores on a discrete, ordinal scale from 0 to 137; lower scores indicate better function.
Time Frame: as for outcome 4
Population: Full Analysis Set: all randomized participants (or parent/proxy) who received at least 1 dose of study drug. Participants who had an assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind UX007 | Double-Blind Placebo
Number analyzed (Participants) | 13 | 15
units on a scale | -2.0 (4.74) | -8.5 (4.41)
Statistical Analysis 1: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.0138, Wilk-Shapiro Test for Normality
Statistical Analysis 2: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Number of participants in this analysis completed both UX007 treatment period and placebo treatment period (n=13); Test type: Superiority; p = 0.3907, Wilcoxon Rank Sum test — [p-value comment as in outcome 4, analysis 1]; Hodges-Lehmann estimate (Median Diff.) = 2.0, 95% CI 2-sided [-3.5 to 20.5]

23. Secondary Outcome: Change From Baseline in CANTAB, Paired Associates Learning First Trial Memory Score (PALFTMS) at Treatment Week 10
Description: CANTAB measures neuropsychological function using a standardized, computerized battery of tests designed to assess visual memory, working memory, new learning and reaction time. PALFTMS assesses the cognitive domain of episodic memory, with scores on a discrete, ordinal scale from 0 to 27; higher scores indicate better function.
Time Frame: as for outcome 4
Population: as for outcome 22
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind UX007 | Double-Blind Placebo
Number analyzed (Participants) | 13 | 15
units on a scale | -0.1 (1.12) | 0.9 (1.04)
Statistical Analysis 1: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.5233, ANCOVA — [p-value comment as in outcome 21, analysis 1]; LS Mean Difference = -1.0, 95% CI 2-sided [-4.4 to 2.4], Standard Error of Mean 1.51
Statistical Analysis 2: Comparison: Double-Blind UX007 vs Double-Blind Placebo; Test type: Superiority; p = 0.6918, Wilk-Shapiro Test for Normality

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 30-35 days after final dose. Mean (SD) treatment duration was 65.7 (12.06) and 68.3 (7.04) days for double-blind UX007 and placebo, respectively, and 305.0 (122.71) days for open-label UX007.
Groups:
- DB UX007: Double-Blind Maintenance Phase: Participants received UX007 (dosed according to an age- and weight-based strategy, up to a maximum daily administration of 130 g) for 10 weeks.
- DB Placebo: Double-Blind Maintenance Phase: Participants received placebo for 10 weeks.
- OL UX007: Open-Label Extension Phase: Participants continued UX007 treatment (dosed according to an age- and weight-based strategy, up to a maximum daily administration of 130 g) for up to 3 years.
Arm/Group | DB UX007 | DB Placebo | OL UX007
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/42 | 0/33
Serious Adverse Events (participants affected / at risk) | 2/43 | 1/42 | 2/33
Other Adverse Events (participants affected / at risk) | 36/43 | 26/42 | 22/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB UX007 (N=43) | DB Placebo (N=42) | OL UX007 (N=33)
Head Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb Asymmetry (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Movement Disorder (Nervous system disorders) | 1 | 0 | 1
Psychomotor Hyperactivity (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB UX007 (N=43) | DB Placebo (N=42) | OL UX007 (N=33)
Abdominal Discomfort (Gastrointestinal disorders) | 4 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 6 | 1 | 5
Abdominal Pain Upper (Gastrointestinal disorders) | 14 | 6 | 7
Anal Incontinence (Gastrointestinal disorders) | 3 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 22 | 5 | 9
Nausea (Gastrointestinal disorders) | 7 | 5 | 4
Vomiting (Gastrointestinal disorders) | 13 | 8 | 8
Fatigue (General disorders) | 3 | 5 | 3
Gait Disturbance (General disorders) | 0 | 1 | 2
Pyrexia (General disorders) | 4 | 1 | 2
Gastroenteritis (Infections and infestations) | 3 | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 0 | 1 | 2
Influenza (Infections and infestations) | 3 | 0 | 2
Viral Upper Respiratory Tract Infection (Infections and infestations) | 5 | 2 | 2
Blood Ketone Body Increased (Investigations) | 3 | 2 | 0
Weight Increased (Investigations) | 3 | 1 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 5 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 2 | 2
Dyskinesia (Nervous system disorders) | 3 | 2 | 3
Headache (Nervous system disorders) | 7 | 6 | 6
Aggression (Psychiatric disorders) | 4 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT02960217/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/17/NCT02960217/SAP_001.pdf